CLINICAL TRIAL: NCT03407339
Title: Shared Oral Care - Improving Oral Care in Institutionalized Elderly in Aalborg
Brief Title: Shared Oral Care - Improving Oral Care in Institutionalized Elderly in Aalborg Municipality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Karin Aagaard, Assistant Professor, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016-899/10-0250
Record Dates: First submitted 2018-01-10; First posted 2018-01-23 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Oral Health; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shared Oral Care Intervention (Active Comparator)
  Interventions: Other: Shared Oral Care intervention
- Control (No Intervention)

INTERVENTIONS:
Other: Shared Oral Care intervention — One hour of teaching in oral hygiene and oral diseases to health care professionals at the intervention nursing homes.
  The dentists will make an assessment of the elderly's oral hygiene at baseline, after three and six months using a mucosal and plaque score. During the six months, a dentist will be doing ward rounds at each nursing home in a specific time interval. In dialog with the resident and the healthcare professional, the dentist will present individual advice on how to perform oral care based on the resident's oral care routines, oral hygiene status, and the resident's physical and cognitive function level.
  Arms: Shared Oral Care Intervention

SUMMARY:
Background:

Nationally and internationally, more people over the age of 65 and especially an increase of people over the age of 80 enter nursing homes with natural dentition and complex prostheses and bridges than previous generations. Furthermore, there is an increased incidence of dental diseases in the elderly. This is leading to increased and different oral care needs. There is a large discrepancy between the elderly who need help with oral hygiene and the elderly who actually receive help. In order to improve the oral hygiene competencies of healthcare professionals at nursing homes, it is necessary to increase their education and improve organizational strategies.

Hypothesis:

The Intervention Shared Oral Care improves the elderlys bleeding and plaque index after 6 months.

Study type:

An intervention study.

A cluster randomization of 14 nursing homes in Aalborg municipality is carried out.

Outcome Measures:

Change in mucosal-plaque score (MPS) index

Change in Oral Related Quality of life

Outcome Measure Time Frame:

Change in mucosal-plaque score index measured at 0, 3 and 6 months.

Change in Oral Related Quality of life measured at 0 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Elderly living in nursing homes in Aalborg Municipality Having one or more natural dentition

Exclusion Criteria:

* no natural dentition

Ages: 65 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 258 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline at 3 and 6 months in MPS index | baseline, 3 and 6 months
  Mucosal Plaque Score Mucosal Score, MS (score 1-4), and Plaque Score, PS (score 1-4). The sum of MS and PS is labeled MI'S (score 2-8). An MPS status is judged as good or acceptable when MI'S = 2-4, as unacceptable when MPS = 5-6, and as poor when MI'S = 7-8.
Change from baseline at 6 months in modified Oral Health Impact Profile (OHIP14) | baseline and 6 months
  modified Oral Health Impact Profile (OHIP14)
  The modified Oral Health Impact Profile:
  1. Have you had painful aching in your mouth?
  2. Do you have trouble biting or chewing any kinds of food, such as firm meat or apples?
  3. Do you limit the kinds or amounts of food you eat because of problems with your dentures?
  4. How often are your teeth or gums sensitive to hot, cold, or sweets?
  Responses are made in a five point scale:
  Very often = 4 Often = 3 Sometimes = 2 Seldom = 1 Never = 0 Do to cognitively impaired elderly the response "I don't know" is added to each question coded 9.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Aagaard, PhD, Principal Investigator — Aalborg University
Locations (1):
- Aalborg University, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No